CLINICAL TRIAL: NCT04609033
Title: Implications of Different Analgesic Models on Inflammatory Markers After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esam Hamed, consultant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17300477
Record Dates: First submitted 2020-09-03; First posted 2020-10-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Perioperative Pain
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Morphine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bupivacaine group (Active Comparator)
  Interventions: Drug: Bupivacaine
- bupivacaine + morphine (Active Comparator)
  Interventions: Drug: Bupivacaine + morphine
- bupivacaine + morphine + ketamine (Active Comparator)
  Interventions: Drug: Bupivacaine + morphine + ketamine
- isotonic saline (Placebo Comparator)
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: Bupivacaine — instillation of local anaesthetic in the abdominal cavity at the end of the procedure
  Arms: bupivacaine group
Drug: isotonic saline — instillation of local anaesthetic in the abdominal cavity at the end of the procedure
  Arms: isotonic saline
Drug: Bupivacaine + morphine — instillation of local anaesthetic + morphine sulfate in the abdominal cavity at the end of the procedure
  Arms: bupivacaine + morphine
Drug: Bupivacaine + morphine + ketamine — instillation of local anaesthetic + morphine sulfate + ketamine in the abdominal cavity at the end of the procedure
  Arms: bupivacaine + morphine + ketamine

SUMMARY:
Postoperative abdominal and shoulder pain that are experienced in patients undergoing laparoscopic cholecystectomy (LC) is significant. Although it is generally less sever than post open cholecystectomy pain, it still causes an avoidable distress in the first 24 hours postoperatively

DETAILED DESCRIPTION:
The incidence of pain after laparoscopy may be as high as 36 to 63 percent and is attributed to the carbon dioxide gas (CO2) used to induce pneumo-peritoneum1.

The residual part of CO2 remains in the peritoneal cavity for several days after the operation and causes stretching of the phrenic nerve endings, local hypothermia, and diaphragmatic irritation by carbonic acid formation

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Laparoscopic cholecystectomy.
* Age spectrum of 18 - 55 years
* ASA I, II
* Have no comorbid chronic medical diseases

Exclusion Criteria:

* Patients with co morbid medical diseases
* Age outside the specified range
* Acute inflammation of the gall bladder
* Critically ill patient
* Emergency operations
* Patient refusal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
postoperative level of ACTH hormone | 6 hours
  a stress marker that increase with pain and surgery

SECONDARY OUTCOMES:
VISUUEAL ANALOGE SCORE | 24 hours
  to assess postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt